PDE4 Inhibition in the Treatment of Seborrheic Dermatitis and Papulopustular Rosacea With PF-07038124

PI: Benjamin Ungar NCT06013371

Document Date: 5/28/2024

#### 

Study ID: STUDY-23-00464 GCO#23-0719

Form Version Date: 2 May 2024

#### **STUDY INFORMATION:**

Study Title: PDE4 Inhibition in the Treatment of Seborrheic Dermatitis and Papulopustular Rosacea With PF-07038124

Study site(s): Icahn School of Medicine at Mount Sinai

Lead Researcher (Principal Investigator): Benjamin Ungar, MD

Physical Address: Icahn School of Medicine at Mount Sinai

Department of Dermatology 5 East 98th Street – 5th Floor

New York, NY 10029

Mailing Address: Icahn School of Medicine at Mount Sinai

One Gustave L. Levy Place - Box 1048

New York, NY 10029

Phone: (212) 241-3288

#### SUMMARY OF THIS RESEARCH STUDY:

This document explains a research study you might be interested in joining. Participation in the study is voluntary. You can agree to join or not. Your decision will not limit your ability to receive care at Mount Sinai. You should only agree to take part if you understand the study and if all of your questions about the research study are answered. If you do join the study, the research team must share any new information with you that may change your mind about taking part.

The purpose of this research study is to evaluate the safety and effectiveness of PF-07038124 in the treatment of seborrheic dermatitis (SD) and papulopustular rosacea (PPR).

If you choose to take part, you will be asked to attend 5 in-person visits over a period of 16 weeks, during which time you cannot participate in another study.

Throughout your study participation the study staff will perform physical examinations, skin assessments, collect blood and urine samples, collect skin samples via non-invasive tape strips, administer questionnaires, and perform urine pregnancy tests (for participants who can possibly get pregnant). There will be no charge to you for your participation in this study. The study drug, study related procedures, and study site visits will be provided at no charge to you or your insurance company.

Data and samples collected during this study will be stored indefinitely.

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



#### 

Study ID: STUDY-23-00464 GCO#23-0719 Form Version Date: 2 May 2024

If you qualify for the study, you will be compensated \$70 for each visit you complete, starting with the Baseline visit (visit #2).

If you choose to take part, the main risks to you are skin irritation (including pimples and skin redness), worsening or no improvement in your SD or PPR.

You may benefit from taking part in this research. Some potential benefits are that the symptoms associated with your SD or PPR may improve.

Instead of taking part in this research, you may seek alternative treatment options which include topical corticosteroids, antifungal creams, antibiotics, acne fighting treatments and or medications that reduce flushing (redness).

If you are interested in learning more about this study, please continue to read below.

#### STUDY PARTICIPATION:

You may qualify to take part in this research study because you are at least 18 years old and have been diagnosed with either mild to moderate seborrheic dermatitis (SD) or papulopustular rosacea (PPR).

Your participation in this research study is expected to last up to 16 weeks.

There are up to 78 people expected to take part in this research study at the Icahn School of Medicine at Mount Sinai.

Funds for conducting this research study are provided by Pfizer, the manufacturer of PF-07038124. The lead researcher/institution are being paid by Pfizer Inc. for the work done for this study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### **DESCRIPTION OF WHAT IS INVOLVED:**

If you agree to take part in this research study, here is what may be involved:

All research visits/activities will be performed at the study site listed on page 1 and will be for research purposes only.

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



### ****


After signing this consent form, we will ask you about your medical history, any medications you are taking, and all prior treatments for your SD/PPR. A research doctor will perform a skin examination to assess your SD/PPR. You will also have a physical examination (including measurement of blood pressure and heart rate) and a urine and blood sample will be collected (approximately 3 ¾ tablespoons blood and 3 teaspoons of urine). The blood sample will include a general blood test as well as a test for hepatitis B, hepatitis C, and human immunodeficiency virus (HIV). These tests must be negative to continue to qualify for the study. A pregnancy test will be performed from the urine collected, if applicable. This test must be negative to continue to qualify for the study.

If you continue to qualify for the study you will return for a baseline visit.

#### Baseline Visit (approximately one hour):

At the Baseline visit you will be asked to complete a questionnaire, the research doctor will perform a skin examination to assess your SD/PPR. You will also have a physical examination (including measurement of blood pressure and heart rate) and a blood sample will be collected (approximately 2 tablespoons). Urine will be collected (2 teaspoons) for a pregnancy test, if applicable. A member of the study team will also collect tiny samples of skin via tape strips. This involves the placement and removal of a series of circular stickers (the size of a quarter) on the most affected area of your face and a non-affected area. Photographs of your left cheek, right cheek and forehead will be taken. All efforts will be made to photograph areas that do not include your eyes or any other identifying markers (tattoos). If there are any views that show your eyes or any identifying markers, they will be blacked out in any publication. You cannot participate in the trial if you do not consent for photographs to be taken.

You will be given your study drug and all subjects will apply the study drug ointment once daily for 8 weeks. Study drug will not be made available to you after the study ends.

You will be asked to return to the study site for additional 3 visits: Week 4, Week 8 (during the treatment period) and at Week 12 (4 weeks after your last application).

#### Weeks 4, 8 and 12 (approximately 1 hour each):

The following procedures will be done at each visit:

- We will ask you about any updates to your medical history and medications you are taking
- You will be asked whether you missed any applications of the study drug (week 4 and 8 only)
- You will be asked to complete a questionnaire
- The research doctor will perform a skin examination to assess your SD/PPR
- You will have a physical examination (including measurement of blood pressure and heart rate)
- Urine will be collected (2 teaspoons) for a pregnancy test, if applicable
- A blood sample will be collected (approximately 2 tablespoons)

-----FOR IRB USE ONLY-----------------------FOR IRB USE ONLY---------------------

Rev 11.11.2022 (Amendment 1-03.09.2023)



#### 


- A member of the study team will also collect tiny samples of skin via tape strips
- Photographs will be taken of both cheeks and forehead (Week 8 and 12 only)
- Blood (2 tablespoons) and urine (2 teaspoons) samples will be collected for standardized tests
- Blood sample (1 tablespoon) will be collected for possible future use.

If you are discontinued or decide to discontinue your participation in this study, you will be asked to return to the site for an Early Termination Visit.

#### Early Termination Visit (approximately 1 hour):

- We will ask you about any updates to your medical history and medications you are taking
- You will be asked whether your missed any applications of the study drug, all study drug will be retrieved
- You will be asked to complete a questionnaire
- The research doctor will perform a skin examination to assess your SD/PPR
- You will have a physical examination (including measurement of blood pressure and heart rate)
- Urine will be collected (2 teaspoons) for a pregnancy test, if applicable
- A member of the study team will also collect tiny samples of skin via tape strips
- Photographs will be taken of both cheeks and forehead
- Blood (2 tablespoons) and urine (2 teaspoons) samples will be collected for standardized tests
- Collect blood sample for possible future mechanistic analyses

Results of the standardized lab tests will be provided to you.

Because this research study involves the use of a study drug, a note must be included in your electronic medical record that you are taking part in the research. This way, anyone involved in your medical care will know that you are a study participant, and they can work to avoid any problems or negative outcomes that could arise if they do not know.

#### Randomization

No one, not you, or anyone from your medical team or from the research team will be able to choose what group you are assigned to or what study drug you get. It will be by chance, like pulling names out of a hat. You will have a 2 in 3 chance of receiving PF-07038124 and 1 in 3 chance of receiving placebo (inactive ointment that looks like PF-07038124). Neither you nor the Lead Researcher or your own doctor will know which study drug you are getting. If there is an emergency, they can get this information.





#### 


#### **HIV/AIDS**

To take part in this research study, your blood will be tested for evidence of HIV, the virus that causes AIDS. People can get HIV through unprotected sexual contact with someone who has HIV, and through contact with blood (as in sharing needles including for piercing, tattooing, and injecting drugs). People who are pregnant with HIV infections can transmit HIV to their infants during pregnancy, delivery or while breastfeeding. There are treatments for HIV/AIDS that can help people stay healthy. People with HIV/AIDS can adopt safe practices to protect uninfected and infected people in their lives from getting HIV or getting infected with a different strain of HIV.

By law, positive test results for HIV/AIDS (as well as other communicable diseases such as hepatitis B, hepatitis C, and syphilis) are reported to the NYS Department of Health so they can study how people get and transmit the disease and notify sexual or needle-sharing partners they may have been exposed. If you wish to be tested anonymously for HIV/AIDS, the research team can refer you to a public testing center, but you will not be able to be in this study. New York State law protects the confidentiality of HIV test results and other related information. It is illegal to discriminate against a person based on their HIV status and services are available to help if this happens. You are free to refuse to get an HIV test, but if you refuse you cannot be part of this research study.

### **Pregnancy**

If you can possibly get pregnant, a urine test for pregnancy will be done before you begin the study and the pregnancy test will be repeated at every visit.

You cannot be included in the study if you are or become pregnant, as the study drug could harm your fetus. You also should not be in the study if you are producing milk to feed a child as the study drug could harm your baby.

Unless you are at least one year past menopause or have had a successful operation to make pregnancy impossible, you should use effective birth control. Unless you are sexually abstinent (not having genital sex) the recommended methods of birth control are:

- The consistent use of approved hormonal birth control (pill, patches, or rings),
- An intrauterine device (IUD)
- Contraceptive injection (Depo-Provera)
- Double barrier methods (Diaphragm with spermicidal gel or condoms (not made of natural membrane) with contraceptive foam)
- Sexual abstinence (no sexual activity)
- Sterilization (a vasectomy, getting tubes tied, or a hysterectomy).

All birth control methods (other than abstinence and sterilization) are only effective if you use them properly, start them at least one month before you begin the research study, and continue using them throughout the research study and for 90 days after the last application of study drug. If you are unsure whether the method of birth control you use is approved to use while you are in this study, you should ask the Lead Researcher before you begin the study. If you are less than one-year post-

Rev 11.11.2022 (Amendment 1-03.09.2023)



### 


menopausal, you could still become pregnant. If you or your partner becomes pregnant, or may be pregnant, at any time during the study, you must tell a person from the research team immediately. The team may stop the study drug and refer you/your partner to an obstetrician/gynecologist for follow-up.

Should you/your partner become pregnant, whether or not you/your partner have the baby, the people funding and overseeing the research may ask for information on the pregnancy, even if you are no longer part of the study. You/your partner will be asked for additional written consent to share this information if that happens.

### Semen/Sperm:

Drugs can be found in semen and alter sperm. Since you are taking part in a study using experimental drugs or treatments, it is recommended that 1) you use a condom, 2) you do not get a partner pregnant or expose them to semen, and 3) you do not donate semen. These recommendations apply both while you are taking the study drug, and for 90 days after you stop taking the study drug. This is because levels of the study drug may be present in the sperm and/or semen even after you stop taking the study drug. You are encouraged to tell your partner(s) and/or their doctor(s) that you are participating in this clinical trial.

#### **USE OF YOUR DATA AND/OR SAMPLES:**

The researchers would like your permission to keep your personal information (such as, name, address, date of birth, social security number), study data and/or samples (blood, tissue, urine) to use or share in future studies. You can still be part of the study if you do not allow us to use or share them. Please select Yes or No to each of the questions below. To decline all future uses/sharing please select 'No' each time. All data and samples will always be linked to your identity, using a code, but that code will always remain with the investigators at Mount Sinai and will not be shared outside of the research team members.

| (1) Will you allow the researchers to store your data and/or samples to use in future research studies? |
|---|
| Please initial your choice: Yes No |
| If you select No, please stop here and move to the next section, 'Your Responsibilities If You Take Part in This Research' section below." |
| If yes, please continue to the next question and tell us how your personal information, study data and/or samples may be used in future research studies. |
| FOR IRB USE ONLY |



### ****


| (2) Do you give the researchers permission to in future studies that are <b>directly related</b> to the | keep the data and/or samples, so they could use them e purpose of the current study? |
|---|---|
| Please initial your choice: YesNo_ | |
| | keep the data and/or samples indefinitely, so they could to the purpose of the current study (for example a |
| Please initial your choice: YesNo_ | |
| and/or samples. This might be in the fields suc | medicine and related sciences would like to use data h as anthropology, human origins, mapping human researchers <b>outside the field of medicine</b> to use your |
| Please initial your choice: YesNo_ | |
| <ul> <li>samples came from you personally, that with the future research in a different area recomples came from, then one of the follow I. If you allowed the researchers to contain explain why your data and/or samples in permission will be asked to use your data. If you do not give permission to be contained in the practical (for example, because you used. The Institutional Review Board (I samples linked to your identity. The IRI identifiable health information without of data and/or samples will not be more the committee of doctors and scientists and</li> </ul> | uires that it is known specifically who the data and/or |
| | and/or samples given <b>to other researchers</b> , including c institutions and for-profit companies, for use in ove? |
| Please initial your choice: YesNo | |
| | 3 USE ONLY |
| Rev 11 11 2022 (Amendment 1-03 09 2023) | |



### 


Whether or not you have allowed us to share your data and/or samples with Pfizer, the researchers at Mount Sinai will keep data and/or samples collected about you during this research study to use in future research studies consistent with the wishes you expressed above.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study, you will be responsible for the following things:

- While you are taking part in this study, you should not take part in another study without notifying the research doctor.
- You must follow the instructions you are given by the research doctor and study staff (including applying the study drug as directed and coming in for all study visits). If you do not follow the instructions, your visit may have to be rescheduled, or you may be discontinued from the study.
- Tell the research doctor or the study staff about all prescription and non-prescription medications, supplements, herbal preparations, or vaccines before you take them.
- Notify the research doctor or study staff if you move and provide your new address and contact information.

#### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

There may be costs to you for taking part in this study. Certain safety tests or assessments may uncover underlying diseases or problems that require medical attention

If you agree to take part in this study, you will be paid \$280 for your time and effort. If you do not complete all visits, then you will be paid \$70 for each visit you complete (Baseline, Week 4, Week 8 and Week 12). Payment will be given to you in the form of a check at the end of the study.

It can take up to 6 weeks to prepare and give you a check for study participation. If you do not get a check by then, you can first contact the research team. If further assistance is needed, please contact Mount Sinai's Program for the Protection of Human Subjects at (212) 824-8200.

Tax law may require the Mount Sinai Finance Department to report the amount of payment you receive from Mount Sinai to the Internal Revenue Service (IRS) or other agencies, as applicable. Generally, this happens if you receive payments that equal \$600 or more from Mount Sinai in a calendar year. You would be responsible for the payment of any tax that may be due.

#### **POSSIBLE BENEFITS:**

There is a chance this study may benefit you, but this is not guaranteed. Others may benefit from what researchers learn from the study. Possible benefits to you include: improvement or clearing of

Rev 11.11.2022 (Amendment 1-03.09.2023)



### 


your SD/PPR symptoms. If this occurs, it would not be permanent. Also, once the study is completed, the study drug will no longer be available to you.

#### **POSSIBLE RISKS AND DISCOMFORTS:**

#### Physical Risks of PF-07038124

Animal studies have been done to understand the potential risks of the study drug in humans. PF-07038124 was studied in rats, dogs, rabbits, and minipigs. When applied on the skin to the minipig as an ointment, redness and swelling of the skin were seen. When given by mouth to rats and dogs, increased heart rate, contractility, and blood pressure were seen. Rats and minipigs also showed injury to blood vessels in the lining of intestine, kidneys, adrenal glands and bladder at non-tolerated doses. Rats, dogs, and minipigs also showed effects on the brain. This included decreased activity, hunched posture, twitching, tremors, and abnormal gait. Effects on the stomach and intestine included vomiting, increased saliva production, and soft stools in rats, dogs, and minipigs. However, animal studies do not always predict the effects people may experience. There are at least two other similar medications, that are both given by mouth. These medications are known to cause injury to blood vessels in animals.

The most commonly reported treatment-related side effect following 10 days of topical application of the PF-07038124 ointment across healthy participants were skin irritation; including pimples and skin redness, which were all reported as mild. There were no treatment-related side effects in the study where PF-07038124 was applied to skin of participants with Atopic Dermatitis and Plaque Psoriasis. A majority of participants had no skin tolerability issues after study treatment application. Of those who did, most cases of skin tolerability issues were mild. There were no cases of pain and itching at the site of application.

The other two similar medications taken by mouth are known to cause nausea, diarrhea, weight loss, headache, difficulty sleeping, anxiety, harming yourself, and depression. Due to expected low system exposure associated with skin administration of PF-07038124, the effects observed with other similar medications taken by mouth are not anticipated.

Another similar topical medication called Crisaborole, is applied on skin to treat eczema. It is known to cause pain and itching at the site of the application.

The study drug, PF-07038124, is applied to the skin. It is not known whether it will have the same side effects as observed with similar medications taken by mouth or applied to the skin.

The effects of PF-07038124 on sperm, a pregnancy, a fetus, or a nursing child are not known. If you are pregnant or become pregnant, this research may hurt your baby or your pregnancy in ways that

-----FOR IRB USE ONLY-------

Rev 11.11.2022 (Amendment 1-03.09.2023)



### 


are unknown. The unknown risks could be minor or major (death) for the pregnancy. You should not become pregnant or get someone pregnant while you take part in this study. Please read the acceptable methods of birth control found under the Description of What Is Involved section of this document.

All drugs have a potential risk of causing an allergic reaction, which (if not treated quickly) could become life-threatening. You or your child should get medical help right away or call your local emergency number and contact the research doctor if you think your child or if your child think they have any of the following symptoms of a serious allergic reaction:Trouble breathing or wheezing; Swelling of the face, mouth, lips, gums, tongue, or neck; Rash, hives, or blisters; Dizziness and fainting; a fast pulse/heart beat; and/or or sweating.

In addition to these risks, this research study may hurt you in ways that are not known. The unknown risks could be minor or major (death).

#### Risk of loss of private information:

This risk always exists, but there are procedures in place to minimize the risk.

#### Risks of Blood Draw:

The risks of a blood draw include pain, bruising, and the slight possibility of infection at the place where the needle goes in. Some people feel dizzy or may faint during or after a blood draw.

### **Group Risks**:

Although your name will not be given to researchers, basic information such as your race, ethnic group, and sex may be shared. This information helps researchers learn whether the factors that lead to health problems are the same in different groups of people. It is possible that such findings could one day help people of the same race, ethnic group, or sex as you. However, they could also be used to support harmful stereotypes or discrimination.

#### Privacy Risks:

Your name and other information that could directly identify you (such as an address, date of birth, or social security number) will never be placed into a database. However, because your genetic information is unique to you, there is a small chance that someone could trace it back to you. The risk of this happening is very small, but may grow in the future. Since the database contains genetic information, a break in security may also pose a potential risk to blood relatives as well as yourself. For example, it could be used to make it harder for you (or a relative) to get or keep a job or insurance. If your private information was misused, it is possible you would experience other harms, such as stress, anxiety, stigmatization, or embarrassment from revealing information about your family relationships, ethnic heritage, or health conditions.



#### 


#### **OTHER OPTIONS TO CONSIDER:**

You may decide not to take part in this research study. If you decide not to take part, this will not affect the clinical care you receive at Mount Sinai. The choice is totally up to you.

Instead of being in this research study, if you have SD your choices may include: topical corticosteroids and antifungal creams. However, they have a maximum duration of use. Using corticosteroids over a long period of time may result in thinning of the skin. If you have PPR your choices may include topical or oral antibiotics, acne fighting treatments, medications that contain sodium sulfacetamide or sulfur, and/or medications that reduce flushing (redness). Taking antibiotics too frequently or for too long can cause a serious health problem called antibiotic resistance. The common risks associated with these other topical treatments include itching, dryness, temporary redness, or irritated skin.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY

If you are injured or made sick from taking part in this study, you will get medical care. The group funding this research study will pay you for any reasonable and necessary medical expenses to diagnose and treat research-related injury or illness. This does not prevent you from seeking payment for injury related to malpractice or negligence. You can contact the Lead Researcher for more information.

The Centers for Medicare and Medicaid Services (CMS) is the government agency that oversees Medicare and Medicaid. Funding agencies who make payments for injuries related to studies must report payments to CMS. In order to do this, the funder must have certain information about you, such as your name, date of birth, Social Security Number, Medicare or Medicaid ID numbers, date of injury, and description of injury. The funding agency is only allowed to use this information to report payments related to the injury should this be necessary or as otherwise specified in the Authorization to Use and Disclose Protected Health Information section, which is included below.

#### **ENDING PARTICIPATION IN THE RESEARCH STUDY:**

You may stop taking part in this study at any time. No matter what you choose, your care and benefits through Mount Sinai will not be negatively impacted.

If you decide to stop being in the study, please contact the Lead Researcher or the research staff. You will be asked to return all study drug and for your safety, you will be asked to complete the Early Termination Visit tests (as described in the description section of this form).

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



#### 

Study ID: STUDY-23-00464 GCO#23-0719

Form Version Date: 2 May 2024

If you decide to stop being in the research study, any improvements in your SD/PPR may be lost or worsen.

You may also withdraw your permission for the researchers to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page. Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you stop being in the research study, the research team may not remove information they have already placed in the study database, and may continue to use that data as part of this study. The research team may ask you whether they can continue to collect information from your medical record. You may inform the study team in writing at any time if you choose to withdraw your consent for future use of any personal information, study data and/or samples.

If you decide you don't want your data and/or samples to be used for research anymore, you can contact the Lead Researcher and ask to have your data and/or samples withdrawn or labeled so that they will not to be used in additional projects or shared. If your data and/or samples have already been shared with researchers, those researchers will be asked to stop using them. However, if any data and/or samples have already been shared without your identity or a linking code, it won't be possible to retrieve them. Data and/or samples that have already been used will not be affected by your decision. If your data and/or samples have already been deposited in an external repository, the study team will request that your data and/or samples be removed.

<u>Withdrawal without your consent</u>: The Lead Researcher, the funder or Mount Sinai may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the research team have not been followed, the Lead Researcher believes it is in your best interest, or for any other reason. If data and/or samples have been stored as part of the research study, they too can be destroyed without your consent.

#### **CONTACT INFORMATION:**

If you have any questions, concerns or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Lead Researcher at phone number 212-241-3288.

If there is an emergency, please call 911 or go to the emergency room. Let the emergency room staff know you are in a research study so they can contact the Lead Researcher if needed.

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



#### 


#### **DISCLOSURE OF FINANCIAL INTERESTS:**

Dr. Benjamin Ungar (the Lead researcher in this study) and Dr. Emma Guttman (a researcher in this study) are paid consultants for Pfizer, the study sponsor and developer of the study drug.

In addition, Dr. Ungar and Dr. Guttman are paid consultants for other companies that research and develop therapies for dermatologic diseases.

If you have questions regarding paid relationships that your physicians/researcher may have with industry, you are encouraged to talk with your physician/researcher, or check for industry relationships posted on individual faculty pages on our website at <a href="http://icahn.mssm.edu/">http://icahn.mssm.edu/</a>.

#### MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:

As part of this study, some of your private and/or protected health information will be obtained, used, and shared with your permission. There is a Federal Health Insurance Portability and Accountability Act (HIPAA) that makes sure this is done correctly and safely.

#### What is protected health information (PHI)?

PHI is the combination of two things:

- 1. PHI contains information that identifies you. It will be used to contact you and link you to your health information, like name, date of birth, medical record number, and address.
- 2. PHI also contains health information, including information about your mental and physical health from your visits to doctors or hospitals, or from study visits.

Every time you visit a hospital or your doctor, PHI is created and recorded in your medical record by your healthcare providers. In the same way, the PHI created as part of this study will be linked to who you are and your medical information.

What PHI is collected and used in this research study, and might also be shared with others? As part of this study, the research team at the hospital(s) involved in the research will collect your name, address, telephone number, birthdate, social security number, and photographic images.

During the study, the researchers will gather information by:

- Reviewing and/or taking your medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- Doing a physical examination that generally also includes blood pressure reading and heart rate.

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



### 


- Completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.
- Reviewing HIV-related information, which includes any information indicating that you have had an HIV-related test, or have HIV infection, HIV-related illness or AIDS, or any information which could indicate that you have been potentially exposed to HIV.

#### Why is your PHI being used?

Researchers need the information that identifies you so they can contact you during the study. They need your health information and the results of any tests and procedures being collected as part of this study to answer the questions posed in the study. The purpose of the study is discussed earlier in this consent form. Before researchers analyze the data, they remove any information that would let others know who you are or that you took part in the study. If researchers publish or present study results at scientific meetings, lectures, or other events, their presentations would not include any information that would let others know who you are, unless you give separate permission to do so.

The Lead Researcher may also use and share the results of these tests and procedures with other healthcare providers at Mount Sinai who are involved in your care or treatment. The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example:

- The Mount Sinai Program for the Protection of Human Subjects is responsible for overseeing research on human participants and may need to see your information.
- If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes.
- If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

#### Who, outside Mount Sinai, might receive your PHI?

As part of the study, the Lead Researcher, research team and others in the Mount Sinai workforce may disclose your PHI, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Lead Researcher.)

- The United States Department of Health and Human Services (DHHS) and the Office of Human Research Protection (OHRP) (the government organization that is responsible for protecting human research participants).
- Our collaborator on this study, Pfizer, Inc., and their representatives or business partners, including those in other countries. Any reference to the collaborator includes their research partners and service provider including companies belonging to the collaborator, and any person or company that acquires them or the rights to the study drug (PF-07038124). The research team will send study data and results to Pfizer. Information sent to Pfizer will not

Rev 11.11.2022 (Amendment 1-03.09.2023)



### 


include information that directly identifies you (such as your name and Social Security number) and will be coded with a participant identification number. In the future, Pfizer and their representatives, may continue to use coded health information that is collected as part of this study. Pfizer may share information from the study with regulatory agencies.

- The United States Food and Drug Administration.

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier, unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Lead Researcher will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board (IRB) allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, OHRP, as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

For how long will Mount Sinai be able to use or disclose your PHI? Your authorization for use of your PHI for this specific study does not expire.

#### Will you be able to access your records?

During your participation in this study, you will not be able to access your medical records. This is done to prevent the knowledge of study results from affecting the reliability of the study. Your information will be available should an emergency arise that would require your treating physician to know this information to best treat you. You will have access to your medical record and any study information that is part of that record when the study is over or earlier, if possible. The research team is not required to release research information to you that is not part of your medical record.

Do you need to give the researchers permission to obtain, use or share your PHI?

NO! If you decide not to let the research team obtain, use or share your PHI, you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment, or enrollment in any health plans or affect your eligibility for benefits.

### 



### 


The research team may ask you whether they can continue to collect information from your medical record. You will also have to decide if you wish to limit the continued use of the information collected during the study. Under US privacy laws you may also withdraw your permission for the researchers to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page.

Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected, but only to complete this research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you have not already received it, you will also be given The Hospital's Notice of Privacy Practices that contains more information about how The Hospital uses and discloses your PHI.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If researchers are reviewing your medical records or asking questions about your medical history or conditions, it is possible that they may learn information related to your HIV status. If that is the case, the following information concerns you. If researchers are not reviewing your medical records or asking questions about your medical history or conditions, then you may ignore the following section.

### **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 416-0197. These agencies are responsible for protecting your rights.

#### How the Institutional Review Board (IRB) can help you:

This research has been reviewed and approved by an Institutional Review Board (IRB). You may reach a representative of the Mount Sinai Program for Protection of Human Subjects at telephone number (212) 824-8200 during regular work hours (Monday-Friday, 9am-5pm, excluding holidays) for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



### 


- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

| FOR IRB USE ONLY |
|------------------|



### 


**ADULT PARTICIPANT:** Your signature below documents your permission to take part in this research study and to the use and disclosure of your protected health information. A signed and dated copy will be given to you. Signature of Participant Printed Name of Participant Date Time PERSON EXPLAINING STUDY AND OBTAINING CONSENT: Signature of Consent Delegate Printed Name of Consent Delegate Date Time **WITNESS SECTION:** My signature below documents that the information in the consent document and any other written information was accurately explained to, and apparently understood by, the participant, and that consent was freely given by the participant. Signature of Witness **Printed Name of Witness** Date Time

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)

